CLINICAL TRIAL: NCT02732236
Title: Hepatitis B Virus Reactivation in Patients With Marginal Zone B-cell Lymphoma After Rituximab Containing Treatment: Consortium for Improving Survival of Lymphoma (CISL) Marginal Zone Lymphoma Cohort Study (MARCO)
Brief Title: Marginal Zone Lymphoma Cohort in Korea
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dong-A University Hospital (Other)
Responsible Party: Principal Investigator, Sung Yong Oh, Associate professor, Dong-A University Hospital
Other Study IDs: CISL-12-07
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Lymphoma, B-Cell, Marginal Zone
Keywords: marginal zone lymphoma; Cohort; Rituximab; HBV
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Rituximab — Cohort observation study

SUMMARY:
Marginal zone lymphoma is a rare of subtype of Non-Hodgkin Lymphoma. Because of its rarity, prospective clinical trial is difficult to conduct. Therefore we want to make prospective MZL patients' cohort for several observation study

DETAILED DESCRIPTION:
Marginal zone lymphoma (MZL) is a distinct subgroup of non-Hodgkin's lymphoma (NHL), which is typically characterized by an indolent clinical course and long survival duration. MZL is responsible for approximately 7~8% of all NHL. In Korea, MZL accounts for 21% of all B-cell lymphoma and is the second most frequent histologic subtype following diffuse large B-cell lymphoma. Annually, an estimated 500 patients are newly diagnosed with MZL. According to the previous large-scale analyses, MZL is usually a quiet indolent malignancy, which generally presents with limited stage of disease. Localized disease may be controlled with local treatment, and a high response rate can be achieved. Advanced MZL is associated with less favorable survival, and appears to be incurable with the currently available therapy. Transformation to large cell aggressive lymphoma may occur in the first recurrence or in subsequent relapses.

Because of its rarity, prospective clinical trial is difficult to conduct. Therefore we want to make prospective MZL patients' cohort for several observation study especially related with Rituximab use (ex, Hepatitis B virus (HBV) reactivation)

ELIGIBILITY:
Inclusion Criteria:

* pathological confirmed marginal zone lymphoma
* No history of chemotherapy
* enable to routine staging w/u and sampling including HBV serology
* informed consent

Exclusion Criteria:

* mixed with other type lymphoma
* refuse informed consent
* co-existing cancer needed treatment
* prior organ transplantation
* accompany with immunodeficiency

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who is diagnosed as a marginal zone lymphoma- nodal MZL, marginal zone lymphoma of MALT type, splenic MZL
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-03; Primary Completion 2020-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Hepatitis B virus reactivation in patients with marginal zone B-cell lymphoma after rituximab containing treatment | up to 12 months
  Rate of HBV reactivation

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Oh, Principal Investigator — Consortium for improving survival of lymphoma office
Locations (1):
- Sung Yong Oh, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Yes
We will share collected data with participated investigators in Korea